CLINICAL TRIAL: NCT03520790
Title: Vitamin D Receptor Agonist Paricalcitol Plus Gemcitabine and Nab-paclitaxel in Patients With Metastatic Pancreatic Cancer
Brief Title: Paricalcitol Plus Gemcitabine and Nab-paclitaxel in Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase II was not pursued due to futility based on the results of the NAPOLI-3 therapeutic clinical trial.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Stand Up To Cancer (Other); Lustgarten Foundation (Other); American Association for Cancer Research (Other)
Responsible Party: Principal Investigator, Kimberly Perez, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-021
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gemcitabine + Nab-paclitaxel + Placebo (Experimental): * Gemcitabine and Nab-paclitaxel is administered intravenously 3 times/cycle.
  * Placebo is administered orally on a daily basis
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Other: Placebo
- Gemcitabine + Nab-paclitaxel + Paricalcitol IV (Experimental): * Gemcitabine + Nab-paclitaxel is administered intravenously 3 times/cycle.
  * Paricalcitol is administered intravenously once weekly.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Paricalcitol
- Gemcitabine + Nab-paclitaxel + Paricalcitol oral (Experimental): * Gemcitabine + Nab-paclitaxel is administered intravenously 3 times/cycle.
  * Paricalcitol is administered orally on a daily basis
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Paricalcitol

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells.
  Other Names: Gemzar
Drug: Nab-paclitaxel — Nab-paclitaxel is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells.
  Other Names: Abraxane
Drug: Paricalcitol — Paricalcitol (IV or oral) is a man-made form of vitamin D. It is thought to work by blocking a signal in the cancer tumor cells that leads to growth and spreading of the tumor.
  Arms: Gemcitabine + Nab-paclitaxel + Paricalcitol IV; Gemcitabine + Nab-paclitaxel + Paricalcitol oral
Other: Placebo — Placebo
  Arms: Gemcitabine + Nab-paclitaxel + Placebo

SUMMARY:
This research study is a two stage study which consists of a safety run-in phase and a randomized phase 2 study which include subjects with previously-untreated, metastatic pancreatic adenocarcinoma. In the run-in safety study, the safety of adding two formulations (IV or Oral) of paricalcitol to a standard chemotherapy program of gemcitabine and nab-paclitaxel will be evaluated. The randomized phase 2 study will evaluate the efficacy of paricalcitol when added to gemcitabine and nab-paclitaxel

The drugs involved in this study are:

* Paricalcitol
* Gemcitabine
* Nab-paclitaxel

DETAILED DESCRIPTION:
Pancreatic cancer is an aggressive disease with treatment options associated with modest benefit, therefore, new treatment options are needed. Paricalcitol is a man-made form of vitamin D. It is thought to work by blocking a signal in the cancer tumor cells that leads to growth and spreading of the tumor. Paricalcitol was approved by the Food and Drug Administration (FDA) for the prevention and treatment of elevated calcium levels associated with chronic renal failure. The FDA has not approved paricalcitol as a treatment for pancreatic cancer. This research study is being performed to evaluate the benefit of paricalcitol in combination with gemcitabine and nab-paclitaxel for this disease.

The FDA (the U.S. Food and Drug Administration) has approved the combination of gemcitabine and nab-paclitaxel as a treatment option for this disease.

Treatment will consists of 4 week treatment cycles. Paricalcitol in the oral formulation will be taken daily, in the intravenous formulation will be administered three times a week. Nab-paclitaxel and gemcitabine will be administered on days 1,8, and 15.

Subjects continue in the study until disease progression, adverse event/toxicity, death or either the subject or sponsor discontinues the study.

In this research study, the main objectives include:

* Assess adverse side effects associated with the combination of paricalcitol with gemcitabine and nab-paclitaxel.
* Evaluate overall survival in patients with pancreatic cancer receiving gemcitabine and nab-paclitaxel with or without paricalcitol.

Phase II was not pursued due to futility based on the results of the NAPOLI-3 therapeutic clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed pancreatic adenocarcinoma or poorly differentiated carcinoma that is metastatic to distant sites.
* Other histologies such as neuroendocrine and acinar cell carcinoma are excluded. Patients with locally advanced, unresectable disease without distant metastases are excluded.
* No prior chemotherapy for locally advanced or metastatic pancreatic cancer.
* Patients are eligible if they received adjuvant treatment after surgical resection with single-agent gemcitabine or gemcitabine plus capecitabine or gemcitabine and nab-paclitaxel or 5-fluorouracil/leucovorin or 5-FU/leucovorin plus irinotecan and oxaliplatin that was completed >12 months before enrollment. Similarly, adjuvant radiation +/- chemosensitization with 5-fluorouracil, capecitabine, or gemcitabine is allowed if completed >12 months before enrollment.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Age greater than or equal to 18 years.
* Patients must have completed any major surgery or open biopsy ≥4 weeks from start of treatment.
* ECOG performance status ≤1 (see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤1.5 × institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Calcium (corrected for albumin) * ≤1 × institutional upper limit of normal
  * Creatinine ≤1.5 × institutional upper limit of normal OR
  * Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × upper limit of normal.
  * Corrected Calcium = serum calcium (mg/dL) + 0.8 (4 - serum albumin (g/dL))
* Ability to understand and the willingness to sign a written informed consent document.
* Negative pregnancy testing for women of child bearing age
* The effects of Paricalcitol, Gemcitabine and nab-Paclitaxel on the developing human fetus are unknown. For this reason and because vitamin D receptor agonist agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment administration

Exclusion Criteria:

* Prior chemotherapy or any other investigational agents for the treatment of locally advanced or metastatic pancreatic cancer
* Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to paricalcitol, gemcitabine or nab-paclitaxel
* Pre-existing hypercalcemia, defined as baseline serum calcium (corrected for albumin) above the institutional upper limit of normal.
* At the time of trial enrollment, vitamin D containing supplements must be stopped and no vitamin D supplements can be taken while the patient is enrolled to the study due to increased risk for hypercalcemia
* At the time of trial enrollment, calcium containing supplements must be stopped and no calcium supplements can be taken while the patient is enrolled to the study due to increased risk for hypercalcemia
* History of symptomatic genitourinary stones (e.g. kidney stones) within the past 12 months
* History of prior or current synchronous malignancy, except:

  * Malignancy that was treated with curative intent and for which there has been no known active disease for >3 years prior to enrollment
  * Curatively treated non-melanoma skin cancer, cervical cancer in situ, or prostatic intraepithelial neoplasia, without evidence of prostate cancer
* Pre-existing, clinically significant peripheral neuropathy, defined as CTCAE grade 2 or higher neurosensory or neuromotor toxicity, regardless of etiology
* Regular use of thiazide diuretics (e.g. hydrochlorothiazide), which can lead to hypercalcemia. Patients must stop these diuretics prior to initiating treatment. Other anti-hypertensive medications can be substituted, as needed.
* Participants receiving any medications or substances that are inhibitors or inducers of CYP450 3A enzyme(s) are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. [see Appendix D]
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant must be able to swallow and absorb pills.
* Pregnant women are excluded from this study because Paricalcitol is a vitamin D receptor agonist agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Paricalcitol, breastfeeding should be discontinued if the mother is treated with Paricalcitol. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Assess adverse events (per CTCAE v4.0 criteria) | 2 years
  Assess the adverse events (per CTCAE v4.0 criteria) associated with the addition of paricalcitol to gemcitabine and nab-paclitaxel in phase I participants.
Overall survival | 2 Years
  Evaluate overall survival (OS) in patients with metastatic pancreatic cancer receiving gemcitabine and nab-paclitaxel with or without paricalcitol in phase I/II participants.

SECONDARY OUTCOMES:
Assess adverse events (per CTCAE v4.0 criteria) | 2 years
  Assess the adverse events (per CTCAE v4.0 criteria) associated with the addition of paricalcitol to gemcitabine and nab-paclitaxel in phase II participants.
Response rate | 2 years
  Determine the number of patients who demonstrated a clinical response assessed by RECIST criteria on imaging to the combination of paricalcitol with gemcitabine and nab-paclitaxel in phase I/II participants.
Progression free survival | 2 years
  Determine the progression free survival derived from the combination of paricalcitol with gemcitabine and nab-paclitaxel in phase I/II participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Perez, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Penn Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No